CLINICAL TRIAL: NCT06771570
Title: Postoperative Pain and Periapical Tissue Healing Following XP-Endo Finisher Activated Silver Nanoparticles Final Irrigation in Necrotic Mandibular Molars. A Randomized Clinical Trial
Brief Title: Postoperative Pain and Periapical Tissue Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radwa fath Ahmed (Other Government)
Responsible Party: Sponsor-Investigator, Radwa fath Ahmed, Assistant Lecturer of Endodontics at Faculty of Dentistry, Deraya University, Faculty of Dental Medicine for Girls
Organization: Faculty of Dental Medicine for Girls (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Necrotic Mandibular Molars
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2022-08

CONDITIONS: Post Operative Pain; Necrotic Mandibular Molars
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): About 16 Persons injected by 5 ml 2.5% NaOCl using conventional Needle Irrigation
  Interventions: Biological: Silver Nanoparticles Irrigation
- Group II (Active Comparator): About 16 Persons injected by 5 ml AgNPs using conventional Needle Irrigation.
  Interventions: Biological: Silver Nanoparticles Irrigation
- Group III (Active Comparator): About 16 Persons injected by 5 ml AgNPs using XP-Endo Finisher activation.
  Interventions: Biological: Silver Nanoparticles Irrigation

INTERVENTIONS:
Biological: Silver Nanoparticles Irrigation — to evaluate the postoperative pain, antimicrobial efficiency, and periapical tissue healing following the use of silver nano particles solution as a final irrigation, using either conventional needle irrigation or XP-Endo Finisher activation, in necrotic mandibular molar teeth.
  Other Names: conventional needle irrigation

SUMMARY:
The success of endodontic treatment derives from the complete elimination of microorganisms capable of causing an intraradicular or extra radicular infection. To achieve a more effective eradication of these microorganisms, endodontic instrumentation must always be implemented with abundant irrigation, which has to achieve chemical, mechanical and biological effects.

The objectives of root canal irrigation are to dissolve vital or necrotic pulp tissues, disrupt endodontic biofilms, neutralize endotoxins and remove the smear layer. Antimicrobial activity and biofilm destruction appear to be the most important objectives targeted towards the etiology of pulp and periradicular infections.

DETAILED DESCRIPTION:
The role of microorganisms in periradicular infection has been well established in endodontic literature, signifying that endodontic treatment will be afflicted with a higher chance of failure if microorganisms persist in the canals at the time of root canal Obturation .

Furthermore, anatomic complexities of the root canals as isthmuses, fins, ramifications, lateral Canals, and dentinal tubules make the situation much more difficult; bacteria harboring such areas become inaccessible to mechanical instrumentation, and protected by tissue residues, dentin, serum and dead cells that inactivate or diminish the efficiency of antimicrobial agents.

Sodium hypochlorite (NaOCl) is regarded as the most potent disinfectant in endodontics due to its excellent ability to dissolve vital and necrotic tissues in addition to its antimicrobial activity. However, intracanal irrigants are only effective when in contact with the surface, and they cannot penetrate deep into the surfaces because of anatomic barriers. NaOCl can penetrate into the dentinal tubules by 130 μm, whereas bacteria can penetrate into the dentinal tubules by 1000 μm.

Silver nanoparticles (AgNPs) can also be used for disinfection because of their optimal antimicrobial properties. They are effective against many microorganisms including E. faecalis . Nanomaterials has dimensions of 1- 100nm, presenting small sizes, large surface/area mass ratio and increased chemical reactivity , the small size of nanoparticles offers a larger surface area for a small volume of the particles. This allows them to exert action even when used in small quantities, the action of AgNPs differ according to size, concentration, and time of application. Moreover, the killing effect of AgNPs against gram-negative and grampositive bacteria increases with decreasing particle size.

Silver nano particles release silver ions which have an electrostatic attraction to sulfur proteins, that results in adherence and disruption of the bacterial membrane, Silver ions can also cause the denaturation of DNA and ribosomes directly. AgNPs can also interrupt signal transduction by dephosphorylation of tyrosine residues on the peptide substrates leading to cell death and apoptosis.

However, cell culture studies revealed that AgNPs are able to induce cytotoxicity in human cell lines including human bronchial epithelial cells, red blood cells, macrophages, liver cells, etc., particularly for those with sizes more than 10 nm, and the cytotoxicity of AgNPs has been reported to be contingent upon dose, size, and exposure time .

Since irrigant needs to reach and disrupt the biofilm matrix in less accessible areas of the root canal system, several agitation and activation methods have been proposed to improve efficacy, including sonic & ultrasonic activation, negative apical pressure irrigation, laser activation and physical agitation using XP-Endo Finisher. Several studies have shown that compared to conventional irrigation, the application of ultrasonic activation or XP-Endo Finisher enhances the efficacy of NaOCl in reducing intra-canal bacteria and removing biofilms from the main canal lumen, the apical third root surface and shallow or deep layers of root dentine.

Pain following root canal treatment is an important patient-centered outcome that has been related to the patient's quality of life, with an incidence of 3-58% following treatment. It could be associated with mechanical and chemical injuries, along with the presence of microorganisms in the periapical region. However, Advancements in material science and metallurgy have improved the predictability and efficiency of delivering endodontic treatment either following single-visit or multiple-visit root canal treatment, even in teeth with necrotic pulps.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Patients between the age group of 20 and 40 years old with no sex predilection, who agree to take partin the study and to sign a written informed consent.
* Asymptomatic necrotic mandibular molars:non-responsive to thermal pulp testing, with no pain to percussion, and distal root having typeI root canal system.
* Presence of periapical radiolucency not exceeding 5mm in diameter,confirmed with cone beam computed tomography scans.

Exclusion Criteria:

* Medically compromised patients, pregnant and lactating females.
* Patients were using medication such as analgesics or any kind of antiinflammatory drugs, or antibiotics 12 h preoperatively.
* Teeth with calcified root canals, external or internal root resorptions, periodontal problems as those with mobility greater than Grade I, or pocket depth exceeding 5 mm.
* Previously endodontically treated teeth, immature with open apex, severe damage and those having associated traumatic occlusion.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Post operative Pain | 4 days
  Following the treatment, patients will be asked to record their pain level on a modified VAS at 4, 24, 48, 72, and 96 h.

SECONDARY OUTCOMES:
Digital periapical radiographs (DPR) | 12 Months
  The patients evaluated by Digital periapical radiographs after irrigation to assess the periapical tissue healing, and confirmed with cone beam computed tomography scans

CONTACTS AND LOCATIONS:
Overall Officials: Wael Hussein Kamel, Professor, Study Chair — Faculty of Dental Medicine for Girls, Al-Azhar University
Locations (1):
- Hospital of Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided